CLINICAL TRIAL: NCT03387748
Title: Role of Semantic Processing and Visuospatial Skills in Production of Iconic Gestures
Brief Title: Cognitive Skills and Iconic Gestures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S61109
Record Dates: First submitted 2017-12-18; First posted 2018-01-02 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Gestures
MeSH Terms: conditions — Gestures

STUDY DESIGN:
Intervention Model Description: non-factorial, cross-sectional study (with control group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gesture elicitation (Experimental): Observation: hand gesture elicitation task
  Interventions: Behavioral: Gesture elicitation

INTERVENTIONS:
Behavioral: Gesture elicitation — * Participants are required to gesture with their hands (and not speaking) one by one 30 pictures from the Boston Naming Task which appear on a laptop screen.
  * Participants retell a cartoon to the researcher
  * The researcher initiates a 10-min spontaneous conversation.
  These three tasks are video-recorded.

SUMMARY:
In this study, cognitive skills will be identified that underlie the production of iconic gestures in individuals with language difficulties. Specifically, what is the role of nonverbal semantic processing and visuospatial skills in the use of iconic gestures?

DETAILED DESCRIPTION:
Individuals with language difficulties (e.g., vocabulary or forming sentences) can find it difficult to communicate and express their thoughts. Speech-language therapists sometimes encourage individuals with language difficulties to use hand gestures. By using gestures these individuals may find it easier to express their thoughts and their communication partners may find it easier to comprehend them. The researchers aim to answer the question: which skills are needed to produce highly comprehensible gestures? The answers to this question can inspire future language therapy for individuals with language difficulties.

Task1. Participants sees 30 items from the Boston Naming Task one by one. The researcher explains that she can not see the screen. When an image appears, the examiner asks the participant to describe the item without speaking, but by using hand gestures. These gesture versions are recorded on video. The researcher indicates which gesture strategy the participant used with each executed gesture (i.e., sketch, shape, object, or deictic). In addition, 200 adults with a typical development assess the intelligibility of each gesture. The recordings are presented one by one in a random order. The evaluators must write down what concept the person depicts on the video. By adding the correct responses per participant, each participant receives a skill score. This skill score is related to the individual results of cognitive testing.

Task2. Participants watch a cartoon. They tell the story to the researcher who "has never seen the cartoon and does not know what is happening". Participants do not receive instructions on the use of gestures. This storytelling task is recorded on video. The researchers will write this down and note which gestures are being produced. The videos are used to calculate two variables: the ratio of the number of gestures to words, and the ratio of gestures that are replacements of speech to all gestures (both speech replacement and complementary to speech). These variables are related to the results of the cognitive tests.

Task3. The researcher starts a 1-on-1 interview (10 minutes) with the participant. This conversation partly proceeds according to a semi-structured script: a few questions have been drawn up in advance. Each question or comment contains two content words that make a gesture possible. During half of the scripted questions, the researcher will not use any gesture. During the other half, the researcher will produce the two gestures. As with a semi-structured interview, the researcher ensures a natural conversation. The conversations are recorded on video. The researcher transcribes the interviews and indicates whether the participant takes over the gestures of the researcher. Each time a script gesture is presented, the examiner indicates whether the participant has responded by applying the spoken word and / or the gesture. By involving the cognitive test results, it can be analyzed whether people with higher semantic processing and higher visual-spatial skills take over from others more often than those with weaker semantic processing skills and weaker visual-spatial skills.

ELIGIBILITY:
Inclusion Criteria:

* Moderate Intellectual disability
* Down syndrome

Exclusion Criteria:

* neurodegenerative disorder
* non-corrected severe hearing impairment
* non-corrected severe visual impairment
* active knowledge of a sign language or manual signing system

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Gesture iconicity | One observation per participant, 2 years to collect data for all participants
  Likert scale score: understandability of each gesture that is performed. Range of each score: 1 (label: not understandable) to 5 (highly understandable) Summed score is used (range 30/150, with 150 highest performance) .

SECONDARY OUTCOMES:
Gesture rate | One testing per participant, over period of 2 years for all participants
  Rate of iconic gestures per word during narrative task
Gesture strategy | One testing per participant, over period of 2 years for all participants
  Rate of iconic gesture strategies: proportion of deictic gestures, proportion of shaping gestures, proportion of handling gestures, and proportion of drawing gestures

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - KULeuven, Leuven, Flanders
  - Katholieke Universiteit Leuven, Leuven, Vlaams-Brabant